CLINICAL TRIAL: NCT06435741
Title: Lymph Node Dissection of Gastric Cancer Based on Molecular Imaging of Metastatic Lymph Nodes of Gastric Cancer with 99mTc-3PRGD2 Probes
Brief Title: Molecular Imaging of Gastric Cancer Metastatic Lymph Nodes with 99mTc-3PRGD2 Probe.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, jiayongning, Doctor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QNJJ2022017
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2023-09

CONDITIONS: Stomach Neoplasm; Lymph Node Metastasis; RADIONUCLIDE IMAGING
Keywords: Gastric cancer; Lymph node metastasis; Tumor molecular imaging; Integrin; Fibroblast activating protein
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): there is only one arm the included patients in which receive 99mTc-3PRGD2 Spect-CT scan.
  Interventions: Diagnostic Test: 99mTc-3PRGD2 Spect-CT scan

INTERVENTIONS:
Diagnostic Test: 99mTc-3PRGD2 Spect-CT scan — Before the operation，SPECT-CT imaging of lymph nodes was performed by integrin αvβ3-specific 99mTc-3PRGD2 probe. The locations of 99mTc-3PRGD2 SPECT-CT were determined by preoperative CT scan. During the operation, D2 lymph node dissection of gastric cancer was performed under the guidance of fluorescent laparoscopy。

SUMMARY:
Surgical lymph node dissection is the key to advanced gastric cancer. In recent years, after the overall implementation of standard D2 dissection, lymph node dissection for gastric cancer began to explore the direction of D1+ again. Current clinical studies of gastric cancer lymph node dissection based on intraoperative fluorescence navigation show that non-tumor specific lymph node fluorescence navigation surgery can only increase the total number of lymph nodes detected and ensure the completion of the dissection but not the accuracy. The sensitivity and specificity of the tracer metastatic lymph nodes are 56.3% (410/728), respectively. Specificity 46.1% (2669/5785). Tumor specific tracing of positive lymph nodes is the key to achieve accurate lymph node dissection for gastric cancer. Although tumor specific tracers are developing rapidly and related clinical studies are gradually being carried out, there are few reports on specific clinical studies on lymph node metastasis, suggesting that lymph node tracing is still a difficult problem. Previous basic studies have suggested that integrins play an important molecular biological role in the process of tumor lymph node metastasis. In the early stage, 99mTc3PRGD2 SPECT-CT showed good lymph node imaging effect in lung cancer and breast cancer, and 99mTc-oncoFAPI PET-CT also showed good lymph node imaging effect in gastric cancer. Therefore, this study aims to explore the application prospect of 99mTc3PRGD2 and other probes in molecular imaging of gastric cancer metastatic lymph nodes and guidance of lymph node dissection and tracer, so as to accumulate preliminary clinical data for exploring corresponding fluorescent probes for intraoperative tracer of gastric cancer lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. Gastric adenocarcinoma was confirmed by histological examination, and the clinical stage was cT2-4N+M0 locally advanced stage;
2. Age 18-75 years old;
3. No previous drug treatment, radiotherapy and other treatments;
4. ECOG 0~1 points, KPS>70 points;
5. The baseline blood routine and biochemical indexes of the subjects meet the following criteria: hemoglobin ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet ≥100×109/L; ALT, AST≤2.5 times the normal upper limit; ALP≤2.5 times the normal upper limit; Serum total bilirubin <1.5 times the normal upper limit; Serum creatinine <1 times the normal upper limit; Serum albumin ≥30g/L;
6. Radical surgical resection (D2 lymph dissection) was performed in all patients.
7. Willing and able to comply with the plan during the study;
8. Provide written informed consent before entering the study screening, and the patient has understood that he or she can withdraw from the study at any time of the study with no loss.

Exclusion Criteria:

1. Pregnant or nursing women;
2. Clinically serious (i.e., active) heart disease, such as symptomatic coronary heart disease, NYHA Class II or worse congestive heart failure, or severe arrhythmia requiring medical intervention (see Appendix 12), or a history of myocardial infarction within the last 12 months;
3. Moderate or severe renal impairment [creatinine clearance equal to or less than 50 ml/min (calculated from Cockroft and Gault equations)], or serum creatinine > the upper limit of normal (ULN);
4. Patients with impaired liver function, ALT or AST less than or equal to 3×ULN, total bilirubin less than or equal to 1.5 ×ULN, or with proven Gilbert syndrome at baseline (unbound hyperbilirubinemia), serum albumin greater than or equal to 3.0 g/dL;
5. History of iodine allergy (ICG contains iodine) or allergy to ICG;
6. History of hyperthyroidism;
7. Under the physiological function state of the general elderly, the drug should be administered with caution.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-06 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 99mTc-3PRGD2 SPECT-CT imaging of metastatic lymph nodes in gastric cancer. | the sensitivity and specificity were determined according to pathological finding after operation.

IPD SHARING:
Plan to Share IPD: No